CLINICAL TRIAL: NCT00779571
Title: Treatment of PCOS (Polycystic Ovary Syndrome)in Morbidly Obese Women - A Randomized Controlled Prospective Dietary Intervention Study
Brief Title: The Female Health Dietary Intervention Study
Acronym: FEMIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Line Kristin Johnson, MSc, PhD, The Hospital of Vestfold
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 86-814d 6.2008.453
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Polycystic Ovary Syndrome; Morbid Obesity
Keywords: Polycystic Ovary Syndrome; Morbid Obesity; Type 2 DM; Coronary heart disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity, Morbid; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crispbread (Experimental): Intervention: Crispbread LCD
  Interventions: Behavioral: Crispbread
- Liquid meal replacement (Active Comparator): Intervention: LMR LCD
  Interventions: Behavioral: Crispbread

INTERVENTIONS:
Behavioral: Crispbread — 8 week low calorie diet

SUMMARY:
This study has two phases:

1. In phase 1 of the study (8 weeks),the effect of two different low calorie diets on manifestations of PCOS, including risk factors for the metabolic syndrome and cardiovascular risk profile will be compared.
2. In phase 2 the long term effect (next 44 weeks) on sustained weight-loss and the above mentioned parameters will be compared and evaluated.

DETAILED DESCRIPTION:
Weight loss is an important and effective treatment of morbidly obese women with PCOS. Effective weight reduction will improve manifestations of PCOS and risk factors for developing type 2 diabetes and coronary heart diseases. We compare the effect of two isocaloric low calorie diets (LCD), - one powder-based shake-diet and a fiber rich diet on the above mentioned parameters. In addition we want to compare the weight-maintenance effect the next 44 weeks of two different follow-up programs: A usual care- and a lifestyle-program.

ELIGIBILITY:
Inclusion Criteria:

* Woman (European Caucasian)
* PCOS
* BMI = or > 35

Exclusion Criteria:

* Cushing syndrome
* Adrenal hyperplasia
* Androgen-producing tumors
* Anovulation caused by hyperprolactinemia
* Pregnancy, breast feeding
* Use of oral contraceptives/hormone treatment/insulin-sensitizing agents

Ages: 19 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | One year

SECONDARY OUTCOMES:
Improvement of PCOS, diabetes type 2- and coronary heart disease-risk factors | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, MD, PhD, Principal Investigator — The Hospital of Vestfold; Tom Tanbo, MD, PhD, Study Chair — Oslo University Hospital; Kirsten B Holven, PhD, Principal Investigator — University of Oslo; Line Kristin Johnson, MSc, Principal Investigator — Oslo University Hospital
Locations (1):
- Kvinneklinikken, Rikshospitalet-Radiumhospitalet HF, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Johnson LK, Holven KB, Nordstrand N, Mellembakken JR, Tanbo T, Hjelmesaeth J. Fructose content of low calorie diets: effect on cardiometabolic risk factors in obese women with polycystic ovarian syndrome: a randomized controlled trial. Endocr Connect. 2015 Sep;4(3):144-54. doi: 10.1530/EC-15-0047. PMID 26138702